CLINICAL TRIAL: NCT02658266
Title: Effect of Resistance Training in Adults With Complex Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GUCHUmU02
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2016-08

CONDITIONS: Congenital Heart Defect
Keywords: resistance training; adult; muscle strength; muscle endurance; muscle metabolism
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): Home based resistance training 12 weeks home based resistance training 3 times per week, 10-12 reps, 2 sets
  Interventions: Behavioral: Home based resistance training
- Control group (No Intervention): No instructed exercise training. Continue with habitual physical activity.

INTERVENTIONS:
Behavioral: Home based resistance training — The participants in the intervention group will receive an individualized resistance training program. The individual adjustments in load will will be made from the results of the muscle function and muscle strength tests. The resistance training will be home based and performed 3 times per week 10-12 reps 2 sets 12 weeks. Increment of load will be performed continuously according to rating of perceived exertion.
  Arms: Resistance training

SUMMARY:
Adults with complex congenital heart disease have impaired muscle function compared both to health controls and patients with lesions classified as simple. There is only one study assessing the effects of resistance training in patients palliated with Fontan procedure. The hypotheses of the present study is that home based resistance training will improve muscle function in adults with different complex congenital hear diseases.

DETAILED DESCRIPTION:
The number of adults with complex congenital heart disease is increasing and today they outnumber the children with corresponding lesions. However, the longterm prognosis is still unknown and continuously changing as new therapeutic options are introduced.

Patients with complex congenital heart disease have reduced muscle function compared to healthy controls as well as patients with lesions classified as simple. Furthermore, men with congenital heart disease are more commonly underweight and less commonly overweight obese compared to the general population. In addition, men with complex lesions are shorter in comparison to controls. This indicates an altered body composition i.e. muscle mass, fat mass and bone density in this population. Moreover, impaired muscle metabolism has been reported in patients palliated with Fontan procedure.

Adult patients with complex congenital heart disease will be recruited based on defined inclusion and exclusion criteria. Muscle function, muscle strength, muscle metabolism and body composition will be evaluated before randomisation and at follow-up after twelve weeks. The patients will be randomised to twelve weeks of home based resistance training or to a control group. The randomisation ratio will be 1:1 ( intervention:control). The control group will be instructed to continue with their habitual physical activities. The resistance training protocol will be individualised based on the results of the muscle function and muscle strength tests.

The aim of this study is to investigate the effects of resistance training on muscle function, muscle strength, body composition and muscle metabolism in adults with complex congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Complex congenital heart disease ( e.g. tetralogy of Fallot, transposition of the great arteries, pulmonary atresia, patients palliated with Fontan procedure or total cavo-pulmonary connection).
* Clinically stable without significant change the last 3 months.
* Adult (> 18 years of age).
* Informed consent.

Exclusion Criteria:

* Cognitive impairment affecting the ability of independent decision making.
* Present strategy of regularly executing resistance training > 2times per week in purpose to increase muscle strength.
* Other comorbidity affecting physical activity.
* Other circumstance making participation unsuitable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength (Newton, N) | Change from baseline muscle strength at 12 weeks follow-up

SECONDARY OUTCOMES:
Change in muscle endurance (number of repetitions) | Change from baseline muscle endurance at 12 weeks follow-up
Change in total body skeletal muscle mass (kg) | Change from baseline total body skeletal muscle mass at 12 weeks follow-up
  Using dual-energy x-ray absorptiometry (DEXA)
Change in appendicular skeletal muscle mass (kg) | Change from baseline appendicular skeletal muscle mass at 12 weeks follow-up
  Using dual-energy x-ray absorptiometry (DEXA)
Change in body fat percentage | Change from baseline body fat percentage at 12 weeks follow-up
  Using dual-energy x-ray absorptiometry (DEXA)
Change in bone mineral density (g/cm2) | Change from baseline bone mineral density at 12 weeks follow-up
  Using dual-energy x-ray absorptiometry (DEXA)
Muscle metabolism | Change from baseline muscle metabolism at 12 weeks follow-up
  near infrared spectroscopy (NIRS)

OTHER OUTCOMES:
Compliance to study protocol | At completion of study protocol 12 weeks
  number of training sessions
Adverse events | Once a week from the date of onset of the home based exercise regimen until the followup at 12 weeks
  Complications to resistance training

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Johansson, MD, Phd, Principal Investigator — Umea University
Locations (3):
- Sweden (3):
  - Skåne University hospital, Lund
  - University Hospital, Umeå
  - University Hospital Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandberg C, Thilen U, Wadell K, Johansson B. Adults with complex congenital heart disease have impaired skeletal muscle function and reduced confidence in performing exercise training. Eur J Prev Cardiol. 2015 Dec;22(12):1523-30. doi: 10.1177/2047487314543076. Epub 2014 Jul 18. PMID 25038081
- [Background] Cordina R, O'Meagher S, Gould H, Rae C, Kemp G, Pasco JA, Celermajer DS, Singh N. Skeletal muscle abnormalities and exercise capacity in adults with a Fontan circulation. Heart. 2013 Oct;99(20):1530-4. doi: 10.1136/heartjnl-2013-304249. Epub 2013 Jul 11. PMID 23846614
- [Background] Kroonstrom LA, Johansson L, Zetterstrom AK, Dellborg M, Eriksson P, Cider A. Muscle function in adults with congenital heart disease. Int J Cardiol. 2014 Jan 1;170(3):358-63. doi: 10.1016/j.ijcard.2013.11.014. Epub 2013 Nov 13. PMID 24295897
- [Background] Sandberg C, Rinnstrom D, Dellborg M, Thilen U, Sorensson P, Nielsen NE, Christersson C, Wadell K, Johansson B. Height, weight and body mass index in adults with congenital heart disease. Int J Cardiol. 2015;187:219-26. doi: 10.1016/j.ijcard.2015.03.153. Epub 2015 Mar 18. PMID 25838217
- [Derived] Williams CA, Wadey C, Pieles G, Stuart G, Taylor RS, Long L. Physical activity interventions for people with congenital heart disease. Cochrane Database Syst Rev. 2020 Oct 28;10(10):CD013400. doi: 10.1002/14651858.CD013400.pub2. PMID 33112424